CLINICAL TRIAL: NCT01545791
Title: A Multicentre, Open Label, Nonrandomised, Non-interventional, Observational, Safety Study in Patients Using Insulin Detemir for the Treatment of Type 1 or Type 2 Diabetes Mellitus: The PREDICTIVE™ Study - Predictable Results and Experience in Diabetes Through Intensification and Control to Target: An International Variability Evaluation
Brief Title: Observational Study to Evaluate the Safety of Levemir® in Patients With Diabetes
Acronym: PREDICTIVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1952
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin detemir users
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Administered once or twice daily depending on patients' needs. Dose adjusted for each patient at the discretion of their treating physician

SUMMARY:
This study is conducted in Europe. The aim of the study is to observe the safety of insulin detemir (Levemir®) in patients with type 1 and type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with type 1 or type 2 diabetes mellitus, including newly diagnosed patients who had never received insulin or an insulin analogue before

Exclusion Criteria:

* Patients whom the physician considered might be noncompliant for any reason; for example, uncooperative attitude, inability to return for the final visit and similar
* Patients previously enrolled in this study
* Patients with a hypersensitivity to insulin detemir

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with type 1 or type 2 diabetes mellitus was eligible for the study, including newly diagnosed patients who had never received insulin or an insulin analogue before
Sampling Method: Non-Probability Sample
Enrollment: 1037 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse drug reactions (SADRs), including major hypoglycaemic events | Weeks 0-26

SECONDARY OUTCOMES:
Number of serious adverse events (SAEs) | Weeks 0-26
Number of all adverse events (AEs) | Weeks 0-26
Number of all hypoglycaemic events | In the 4 weeks preceeding week 26
Weight change | Week 0, week 26
Glycosylated haemoglobin (HbA1c) | Week 26
Variability in fasting plasma glucose (FPG) | Week 26
Average plasma glucose level | Week 26
Quality of Life as assessed by a treatment satisfaction questionnaire | Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, London, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com